CLINICAL TRIAL: NCT04844892
Title: A Protocol Investigating the Impact of Lungpacer PROTECT Diaphragm Pacing Therapy on Gas Exchange, Hemodynamics, Regional Lung Ventilation and Atelectasis in Patients Presenting With Moderate ARDS
Brief Title: Phrenic Nerve Stimulation-Induced Lung ReAeration Trial
Acronym: PIRAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-400
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilation Therapy; Complications
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROTECT Diaphragm Pacing Therapy (Experimental)
  Interventions: Device: Lungpacer PROTECT Diaphragm Pacing Therapy

INTERVENTIONS:
Device: Lungpacer PROTECT Diaphragm Pacing Therapy — PROTECT diaphragm pacing therapy is intended to stimulate the diaphragm to preserve and improve inspiratory muscle strength in mechanically ventilated patients.
  Other Names: Lungpacer PROTECT DPTS

SUMMARY:
The Lungpacer PROTECT Diaphragm Pacing Therapy System (DPTS) is a temporary, percutaneously-placed, transvenous, phrenic nerve-stimulating device intended to stimulate the diaphragm to preserve and improve inspiratory muscle strength in mechanically ventilated patients. The purpose of the PROTECT DPTS is to improve gas exchange, regional lung ventilation, and hemodynamics, and decrease atelectasis in patients presenting with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
The PIRAT clinical study is intended to assess the feasibility, safety and effectiveness of transvenous phrenic-nerve-stimulating diaphragm pacing on clinical outcomes in mechanically ventilated patients. By delivering electrical stimulation to the phrenic nerves, which in turn causes the diaphragm muscle to contract, the PROTECT DPTS is intended to protect the diaphragm from atrophy and preserve lung mechanics to reduce lung inflammation and injury associated with short-term mechanical ventilation. Sustained lung and diaphragm health during early mechanical ventilation is expected to reduce the risk of comorbidities, improve clinical outcomes such as weaning success, and thereby reduce the number of patients who require prolonged mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older
* Have been mechanically ventilated due to moderate ARDS for 48-120h
* Have a PaO2/FiO2 ratio < 200 and > 100 at the time of screening with PEEP ≥ 5 cmH2O
* Are expected to remain on mechanical ventilation ≥ 48 hours
* Are under continuous sedation with Richmond Agitation Sedation Scale (RASS) ≤ -3

Exclusion Criteria:

* Septic shock with hemodynamic instability (norepinephrine or epinephrine < 0.5 gamma/kg/min)
* Catheter access to left subclavian vein deemed impossible
* Use of neuromuscular blocking agents within last 12 hours
* Bacteremia within the last 48 hours or uncontrolled source of infection
* Currently on ECMO
* Enrolled in any other study of an investigational drug or device, which may affect the outcomes of the current study
* Pre-existing neurological, neuromuscular or muscular disorder that could affect the respiratory muscles
* BMI >45 kg/m2
* Known or suspected phrenic nerve paralysis
* Any electrical device (implanted or external) that may be prone to interaction with or interference from the Lungpacer PROTECT DPTS, including neurological pacing/stimulator devices and cardiac pacemakers and defibrillators
* No affiliation to the French health insurance system
* Under curatorship
* Imprisoned
* Known or suspected to be pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Changes in PaO2/FiO2 ratio | Day 1
  The changes in PaO2/FiO2 ratio during each acute standard of care ventilation and acute PROTECT pacing therapy session.

SECONDARY OUTCOMES:
Successful LIVE catheter placement | Day 1
  LIVE Catheter was successfully inserted into the left subclavian vein, positioned in accordance with the LIVE Catheter IFU, and the diaphragm was stimulated.
Alveolar-arterial (A-a) gradient | Day 1
  Alveolar-arterial (A-a) gradient documenting gas exchange during each acute standard of care ventilation and acute PROTECT pacing therapy session.
Cardiac output index | Day 1
  Pulse contour cardiac output index assessed by transpulmonary thermodilution during each acute standard of care ventilation and acute PROTECT pacing therapy session.
Regional lung ventilation | Day 1
  Regional lung ventilation assessed using electrical impedance tomography during each acute standard of care ventilation and acute PROTECT pacing therapy session.
Regional lung atelectasis | Day 1
  Regional lung atelectasis assessed using electrical impedance tomography during each acute standard of care ventilation and acute PROTECT pacing therapy session.
Serious adverse events | Day 5
  Occurrence of pneumothorax, significant bleeding and desaturation serious adverse events.

OTHER OUTCOMES:
Days until successful weaning | Day 5
Mortality | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dres, MD, Principal Investigator — AP-HP Hôpital La Pitié-Salpêtrière
Locations (1):
- Hôpital La Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No